CLINICAL TRIAL: NCT01355809
Title: Single Centre, Exploratory, Phase II, Cross-over, Randomised Trial, Evaluating the Effect of Spontaneously Breathing He/O2 65%/35% to Either Spontaneously Breathing N2/O2 65%35% or Non-Invasive Ventilated N2/O2 65%/35% on a 6 Minute Walk Test in Severe COPD Patients
Brief Title: Six-Minute Walk Test Comparing Helium/Oxygen to Nitrogen/Oxygen for COPD Rehabilitation
Acronym: rehabilitate
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to low recruitment rate the sponsor decided to discontinue the study.
Sponsor: Air Liquide SA (Industry)
Collaborators: Asklepios Kliniken Hamburg GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALMED-07-C2-017
Record Dates: First submitted 2011-05-17; First posted 2011-05-18 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Six-Minute Walk Test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Inhalation Nitrogen/Oxygen (Active Comparator): Nitrogen/Oxygen (65%/35%)
  Interventions: Drug: Inhalation Nitrogen/Oxygen
- Inhalation Helium/Oxygen (Experimental): Helium/Oxygen (65%/35%)
  Interventions: Drug: Inhalation Helium/Oxygen
- Inhalation gas (Experimental): Medicinal oxygen 100% via NIV with FiO2 of 0.35
  Interventions: Drug: Inhalation gas

INTERVENTIONS:
Drug: Inhalation gas — Inhalated gas, medicinal oxygen 100% via NIV with Fi O2 0.35, one time by random, 6 minutes
  Other Names: Experimental
  Arms: Inhalation gas
Drug: Inhalation Nitrogen/Oxygen — Inhalated gas, Nitrogen/Oxygen (65%/35%), one time by random, 6 minutes
  Other Names: Active Comparator
  Arms: Inhalation Nitrogen/Oxygen
Drug: Inhalation Helium/Oxygen — Inhalated gas, Helium/Oxygen (65%/35%) one time by random, 6 minutes
  Other Names: Experimental He
  Arms: Inhalation Helium/Oxygen

SUMMARY:
The purpose of this study is to evaluate effects of inspired gas mixtures on the distance walked by patients with severe Chronic Obstructive Pulmonary Disease (COPD) during a Six-Minute Walk test.

DETAILED DESCRIPTION:
the purpose of this study is to evaluate the distance walked by patients with severe Chronic Obstructive Pulmonary Disease (COPD) during a Six-Minute Walk test (6MWT) while breathing Helium/Oxygen 65%/35% compared to either breathing Nitrogen/Oxygen 65%/35% or receiving Non-Invasive Ventilation (NIV) with a FiO2 of 0.35 and to evaluate exercise related symptoms

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged >= 45 and <= 75 years old
* Patient with documented clinical diagnosis of stage III/IV COPD
* Patient with stable COPD defined by no significant increase in COPD medication, no treatment for COPD in an emergency, no acute intensive care setting and no intake of antibiotics in the four weeks prior to selection

Exclusion Criteria:

* Inability or contra-indication to perform pulmonary function tests
* Inability or contra-indication to perform the 6MWT with a trolley
* Any contra-indication to receive NIV
* Obese patient having a Body Mass Index (BMI) > 35
* Pregnant or lactating woman
* Female or chil-bearing potential with lack of efficient contraception

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Distance walked | 6 minutes
  evaluate the distance walked by patients during a Six-Minute Walk Test

SECONDARY OUTCOMES:
Assessment of the safety of inhalation Helium/Oxygen | 6 minutes
  evaluate the safety of the administration of Helium/Oxygen 65%/35%

CONTACTS AND LOCATIONS:
Overall Officials: Karl HAUSSINGER, Prof Dr Med, Principal Investigator — Asklepios fachkliniken München-Gauting
Locations (1):
- Asklepios Fachkliniken München-Gauting, Gauting, Gauting, Germany